CLINICAL TRIAL: NCT04755439
Title: Evaluation of Cerebral Parenchymal Changes in Patients Undergoing Proximal Aortic Surgery With Deep Hypothermic Circulatory Arrest Using Diffusion MR
Brief Title: Evaluation of Cerebral Parenchymal Changes in Patients Undergoing Proximal Aortic Surgery With Deep Hypothermic Circulatory Arrest Using Diffusion MRI
Acronym: NON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Burak Bozkurt, Principal Investigator,, Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/KK / 239
Record Dates: First submitted 2021-01-28; First posted 2021-02-16 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Infarct; Neurological Morbidity; Neurological Complication
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Intervention Model Description: Single center prospective clinical research
Masking Description: non
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- undergoing deep hypothermic cırculatory arrest patients (Other): Difüsıon magnetic rezonans imaging , neuron spesific enolase enzym level , deep hypotermic cırculatory arrest
  Interventions: Procedure: DHCA

INTERVENTIONS:
Procedure: DHCA — DHCA THE USE OF SEREBRAL PROTECTİON TECHNİQUE

SUMMARY:
Deep hypothermic circulatory arrest (DHCA) (18 degree) without cerebral perfusion is a safe technique. Resarchers use this technique in patients with proximal aortic pathologies.

During the DHCA period, cerebral silent ischemic events may occur. But the silent ischemic events don't neurological problems with patients.

DETAILED DESCRIPTION:
It is important to evaluate neurological functions in patients with ascending aortic and aortic root aneurysms who underwent deep hypothermic circulatory arrest (18 degrees) and did not undergo cerebral perfusion. However, neurological changes that are reflected in the clinic are not always encountered. Using preoperative and postoperative diffusion magnetic resonance imaging, silent ischemic lesions that are not reflected in the clinic can be detected. Although there are studies using DW-MRI in patients undergoing different cerebral protection methods in the literature, there are no studies conducted on patients who underwent deep hypothermic circulatory arrest without cerebral perfusion.

To detect silent ischemic lesions with preoperative and postoperative diffusion magnetic resonance method in patients with ascending aortic and aortic root aneurysms undergoing deep hypothermic circulatory arrest (18 degrees) and without cerebral perfusion, and to investigate the correlation between preoperative and postoperative neuron-specific enolase levels and serbral findings.

Cerebral ischemic lesions that may occur in patients undergoing deep hypothermic circulatory arrest (18 degrees) and undergoing ascending aortic and aortic root aneurysm surgery without cerebral perfusion will be detected, and the clinical follow-up and treatment of the patients will be better managed.

We base the imaging of diffusion MR among the examinations to be performed on literature studies that show that withdrawal of patients in the early postoperative period (3rd-7th days) due to the surgical method to be performed without cerebral perfusion under deep hypothermic circulatory arrest, increases the specificity and sensitivity of the test. Therefore, the application of diffusion MR imaging in the early postoperative period (3rd-7th days) after a surgical technique performed under deep hypothermic circulatory arrest (18 degrees) without cerebral perfusion constitutes an indication for diffusion MR in order to detect cerebral ischemic lesions in the early period. Therefore, diffusion MR imaging to be taken in the early period (3rd-7th days) will provide us with the opportunity to create an effective algorithm in terms of patient treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ascending aorta and aortic root aneurysm.
* 18-85 years old

Exclusion Criteria:

* Patients without ascending aortic and aortic root aneurysms
* outside the age range of 18-85, emergency surgery,
* Exceeding the magnetic resonance imaging extraction time limit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Measuring postoperative changes in cranial diffusion MR imaging. | Preoperative (1-3 days before operation time) and postoperative (until the 7th day) cranial diffusion MR of the patients will be taken and compared
  Changes due to new ischemia or hypoperfusion in the cerebral and cerebellar hemispheres will be measured in terms of volume(cm square or mm square). The measurements will be determined using cranial diffusion mr.

SECONDARY OUTCOMES:
the comparison of the preoperative and postoperative neuron spesific enolase enzyms level. | The neuron-specific enolase levels of the patients will be checked in the morning of the operation and postoperatively (up to 6-36 hours).
  The neuron-specific enolase levels of the patients will be checked in the morning of the operation and postoperatively (until 6-36 hours). Neuron-specific enolase enzyme levels will be measured from the blood sample.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kaplan, Prof. Dr, Principal Investigator — Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Locations (1):
- Dr. Siyami Ersek Thoracic And Cardiovascular Surgery Training And Research Hospital., Istanbul, Üsküdar/ Selimiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
starting 6 months after publication).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication).
Access Criteria: Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code